CLINICAL TRIAL: NCT00804908
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Evaluating the Efficacy of ABT-888 in Combination With Temozolomide Versus Temozolomide Alone in Subjects With Metastatic Melanoma
Brief Title: A Study Evaluating Efficacy of ABT-888 in Combination With Temozolomide in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-440; 2008-004941-27 (EudraCT Number)
Record Dates: First submitted 2008-12-01; First posted 2008-12-09 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-03

CONDITIONS: Melanoma; Metastatic Melanoma; Skin Cancer
Keywords: Temozolomide; Skin cancer; Melanoma; Metastatic Melanoma; ABT-888; MM
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Temozolomide; veliparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo for ABT-888 BID + TMZ QD (Placebo Comparator): Placebo for ABT-888 twice daily (BID) for 7 days every 28 days plus temozolomide (TMZ; by body surface area) 150 mg/m2 once daily (QD) for 5 days every 28 days.
  Interventions: Drug: temozolomide; Other: Placebo
- ABT-888 20 mg BID + TMZ QD (Active Comparator): ABT-888 20 mg twice daily (BID) for 7 days every 28 days plus temozolomide (TMZ; by body surface area) 150 mg/m2 once daily (QD) for 5 days every 28 days.
  Interventions: Drug: temozolomide; Drug: ABT-888
- ABT-888 40 mg BID + TMZ QD (Active Comparator): ABT-888 40 mg twice daily (BID) for 7 days every 28 days plus temozolomide (TMZ; by body surface area) 150 mg/m2 once daily (QD) for 5 days every 28 days.
  Interventions: Drug: temozolomide; Drug: ABT-888

INTERVENTIONS:
Drug: temozolomide — temozolomide capsule administered orally once daily for 5 days every 28 days
  Other Names: Temodar; Temodal
Drug: ABT-888 — ABT-888 capsule administered orally twice daily for 7 days every 28 days
  Other Names: veliparib
  Arms: ABT-888 20 mg BID + TMZ QD; ABT-888 40 mg BID + TMZ QD
Other: Placebo — Placebo for ABT-888 capsule administered orally twice daily for 7 days every 28 days
  Arms: Placebo for ABT-888 BID + TMZ QD

SUMMARY:
The purpose of this study is to evaluate the efficacy of ABT-888 in combination with temozolomide versus temozolomide alone in subjects with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (or cytologically) confirmed metastatic melanoma.
* Unresectable Stage III or Stage IV metastatic melanoma.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Subjects with no history of brain metastases demonstrated by a baseline MRI, or subjects with a history of previously treated brain metastases who have history of operable/SRS treatable brain metastases and completed surgical resection/stereotactic radiosurgery with or without adjuvant whole brain radiation at least 28 days prior to Day 1; have baseline MRI that shows no evidence of active intercranial disease; have discontinued taking medications for symptom management of brain metastases at least 7 days prior to Day 1
* 28 days since prior anti-cancer therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* Adequate hematologic, renal and hepatic function.
* Partial Thromboplastin Time (PTT) is <= 1.5 x upper normal limit of institution's normal range and international normalized ratio (INR) < 1.5.
* Subject's with significant fluid retention may be allowed at the discretion of the investigator.
* Life expectancy > 12 weeks.
* Females must not be pregnant.
* Voluntarily signed informed consent.

Exclusion Criteria:

* Lactate Dehydrogenase (LDH) > 2 x Upper Limit of Normal (ULN).
* Ocular malignant melanoma.
* History of central nervous system metastases or leptomeningeal disease.
* Prior treatment with Dacarbazine (DTIC) or Temozolomide (TMZ).
* Prior DNA damaging agents or cytotoxic chemotherapy.
* Prior Whole Brain Radiation Therapy (with exceptions).
* Received an investigational agent within 28 days of study.
* History of seizure disorder and/or taking medication for seizure disorder.
* Active malignancy within the past 5 years, except cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.
* Medical condition that would cause a high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2009-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Result] Middleton MR, Friedlander P, Hamid O, Daud A, Plummer R, Falotico N, Chyla B, Jiang F, McKeegan E, Mostafa NM, Zhu M, Qian J, McKee M, Luo Y, Giranda VL, McArthur GA. Randomized phase II study evaluating veliparib (ABT-888) with temozolomide in patients with metastatic melanoma. Ann Oncol. 2015 Oct;26(10):2173-9. doi: 10.1093/annonc/mdv308. Epub 2015 Jul 22. PMID 26202595

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 346 subjects were randomized; 2 subjects did not receive study drug and were excluded from the safety analysis.
Period: Overall Study
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Started (Intent-to-treat (ITT) population defined as all randomized subjects.) | 115 | 116 | 115
Completed | 0 | 0 | 1
Not Completed | 115 | 116 | 114
Not completed — Other | 115 | 116 | 114

BASELINE CHARACTERISTICS:
Population: ITT population defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD | Total
Number analyzed (Participants) | 115 | 116 | 115 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.13) | 58.6 (12.55) | 62.3 (13.50) | 59.8 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 45 | 38 | 119
  Male | 79 | 71 | 77 | 227

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Time to Event
Description: PFS: the number of days from the date that the participant was randomized to the date the participant experienced a confirmed event of disease progression (radiological, as determined by the central imaging center; or clinical, as determined by the investigator), or to the date of death (all causes of mortality) if disease progression was not reached. All events were included whether the participant was still taking or had discontinued study drug. Events of death were included for participants who had not experienced a confirmed event of disease progression, provided the death occurred within 8 weeks of the last available disease progression assessment. The distribution of PFS, as determined by the central imaging center (radiological)/ investigator (clinical), was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% confidence intervals (95% CIs) for the quartiles for the PFS distribution are provided.
Time Frame: Every Cycle (28 Days) until disease progression was observed or another reason for discontinuation of assessments was identified by the investigator. The maximum observed followup duration at the progression-free survival analysis time was 9.7 months.
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
days
  25th Percentile | 54 [50 to 56] | 56 [53 to 58] | 53 [51 to 56]
  50th Percentile | 60 [57 to 111] | 113 [92 to 168] | 110 [57 to 125]
  75th Percentile | 163 [113 to 283] | 225 [169 to NA] — NA=Not calculable due to insufficient progression events | 226 [173 to NA] — NA=Not calculable due to insufficient progression events
Statistical Analysis 1: Comparison: Placebo for ABT-888 BID + TMZ QD vs ABT-888 20 mg BID + TMZ QD; Comparisons between treatment groups were performed using a Comparisons between treatment groups were performed using a log-rank test stratified by baseline lactate dehydrogenase (LDH) status (0 to 1 ULN; >1 to ≤ 2 ULN) and history of previously treated brain metastases (with, without). Hochberg testing procedure for multiplicity adjustment; Test type: Superiority or Other; p = 0.071, Stratified log-rank
Statistical Analysis 2: Comparison: Placebo for ABT-888 BID + TMZ QD vs ABT-888 40 mg BID + TMZ QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.233, Stratified log-rank

2. Secondary Outcome: Overall Survival (OS): Time to Event
Description: OS was defined as the number of days from the date the participant was randomized to the date of death. All deaths were included, whether the participant was still taking or had discontinued study drug. If a participant had not died and was lost to follow-up, then data were censored at the last study visit or contact date, or date the participant was last known to be alive, whichever was later; if the participant was not lost to follow-up, then data were censored at the last study visit or contact date, whichever was later. The distribution of OS was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% CIs for the quartiles for the OS distribution are provided. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ groups were statistically significantly better than the Placebo + TMZ group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints.
Time Frame: Per protocol, survival follow-up information was to be obtained every 3 months for up to 18 months after the final visit for the subject. The maximum observed follow-up at the overall survival analysis time was 21.0 months.
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
days
  25th Percentile | 207 [155 to 241] | 204 [175 to 247] | 181 [154 to 266]
  50th percentile | 390 [299 to 436] | 327 [274 to 399] | 412 [346 to 483]
  75th percentile | 559 [476 to 598] | NA [492 to NA] — NA=Not calculable due to insufficient survival events | NA [NA to NA] — NA=Not calculable due to insufficient survival events

3. Secondary Outcome: 12-Month Overall Survival (OS) Rate
Description: The 12-month overall survival rate was defined as the percentage of participants surviving at 12 months. The distribution of 12-month OS rate was estimated using Kaplan-Meier methodology. Point estimates and 95% CIs for the quartiles for the PFS distribution are provided. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ treatment groups were statistically significantly better than the Placebo + TMZ treatment group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: Per protocol, survival was to be assessed every 4 weeks or as needed after participant is registered as off-study for up to 18 months. The maximum observed follow-up at the overall survival analysis time was 21.0 months.
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
percentage of participants | 52.6 [43.1 to 61.3] | 43.5 [34.3 to 52.3] | 54.1 [44.5 to 62.7]

4. Secondary Outcome: 6-month Progression-Free Survival Rate
Description: The 6-month progression-free survival rate was defined as the percentage of participants without disease progression at 6 months.The distribution of 6-month progression-free survival rate, as determined by the central imaging center (radiological)/ investigator (clinical), was estimated using Kaplan-Meier methodology. Point estimates and 95% CIs for the quartiles for the PFS distribution are provided. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ treatment groups were statistically significantly better than the Placebo + TMZ treatment group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: as for outcome 1
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
percentage of participants | 19.1 [10.9 to 29.0] | 32.8 [22.0 to 44.1] | 30.7 [20.3 to 41.7]

5. Secondary Outcome: Objective Response Rate
Description: The objective response rate was defined as the percentage of participants with a confirmed CR or PR per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by computed tomography (CT) scan: complete response (CR), disappearance of all target lesions; partial response (PR), ≥30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ treatment groups were statistically significantly better than the Placebo + TMZ treatment group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: Every 2 cycles (8 weeks) until disease progression was observed or another reason for discontinuation of assessments was identified by the investigator. The maximum observed followup duration at the progression-free survival analysis time was 9.7 months.
Population: All subjects in the ITT population (defined as all randomized participants) with measurable disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
percentage of participants | 7.0 [3.1 to 13.2] | 10.3 [5.5 to 17.4] | 9.6 [4.9 to 16.5]

6. Secondary Outcome: Time to Disease Progression
Description: The distribution of time to disease progression, as determined by the central imaging center (radiological)/ investigator (clinical), was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% CIs for the quartiles for the PFS distribution are provided. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ treatment groups were statistically significantly better than the Placebo + TMZ treatment group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: Every Cycle (28 Days), until disease progression was observed or another reason for discontinuation of assessments was identified by the investigator. The maximum observed followup duration at the progression-free survival analysis time was 9.7 months.
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
days
  25th Percentile | 54 [50 to 56] | 56 [53 to 57] | 53 [51 to 56]
  50th percentile | 60 [57 to 111] | 113 [92 to 168] | 110 [57 to 125]
  75th percentile | 163 [113 to 283] | 225 [169 to NA] — NA=Not calculable due to insufficient progression events | 226 [173 to NA] — NA=Not calculable due to insufficient progression events

7. Secondary Outcome: Disease Control Rate
Description: The disease control rate was defined as the percentage of participants who had at least stable disease (complete response, partial response, or stable disease) through the end of Week 8. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ treatment groups were statistically significantly better than the Placebo + TMZ treatment group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: Week 8
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
percentage of participants | 48.7 [39.3 to 58.2] | 62.9 [53.5 to 71.7] | 59.1 [49.6 to 68.2]

8. Secondary Outcome: Time to Neurological/Brain Metastases Progression
Description: Time to neurological/brain metastases progression, defined as the number of days from the date of randomization to the date the participant experienced an event of neurological/brain metastases progression, was estimated using Kaplan-Meier methodology. Point estimates and 95% CIs for the quartiles for the distribution are provided. All events of progression were included, regardless of whether the event occurred while the participant was still taking study drug. If a participant did not experience an event, data were censored at the date of the last available brain CT scan. For participants with no postbaseline brain CT scans, data were censored at randomization. Per protocol, because neither the ABT-888 20 mg BID + TMZ nor ABT-888 40 mg BID + TMZ groups were statistically significantly better than the Placebo + TMZ group for the primary endpoint of PFS, confirmatory statistical testing was not continued for any secondary endpoints, regardless of the observed P values.
Time Frame: as for outcome 5
Population: ITT population defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Number analyzed (Participants) | 115 | 116 | 115
days
  25th Percentile | 60 [34 to NA] — NA=Not calculable due to insufficient progression events | 119 [48 to NA] — NA=Not calculable due to insufficient progression events | 184 [51 to NA] — NA=Not calculable due to insufficient progression events
  50th percentile | NA [60 to NA] — NA=Not calculable due to insufficient progression events | NA [119 to NA] — NA=Not calculable due to insufficient progression events | 184 [184 to NA] — NA=Not calculable due to insufficient progression events
  75th percentile | NA [NA to NA] — NA=Not calculable due to insufficient progression events | NA [119 to NA] — NA=Not calculable due to insufficient progression events | NA [184 to NA] — NA=Not calculable due to insufficient progression events

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 5.6 years); SAEs were collected from the time informed consent was obtained (up to 5.7 years).
Arm/Group | Placebo for ABT-888 BID + TMZ QD | ABT-888 20 mg BID + TMZ QD | ABT-888 40 mg BID + TMZ QD
Serious Adverse Events (participants affected / at risk) | 28/113 | 27/116 | 31/115
Other Adverse Events (participants affected / at risk) | 112/113 | 116/116 | 113/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for ABT-888 BID + TMZ QD (N=113) | ABT-888 20 mg BID + TMZ QD (N=116) | ABT-888 40 mg BID + TMZ QD (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 3
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 3
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 3 | 4
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 2 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1
MELAENA (Gastrointestinal disorders) | 0 | 0 | 1
MOUTH SWELLING (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 1 | 1
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 2 | 1
DEATH (General disorders) | 0 | 1 | 0
DISEASE PROGRESSION (General disorders) | 2 | 0 | 1
FATIGUE (General disorders) | 1 | 0 | 0
PAIN (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 1 | 1
CHOLANGITIS (Hepatobiliary disorders) | 0 | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
GLIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
APHASIA (Nervous system disorders) | 1 | 0 | 0
ATAXIA (Nervous system disorders) | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
TREMOR (Nervous system disorders) | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 0
URETHRAL PROLAPSE (Renal and urinary disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for ABT-888 BID + TMZ QD (N=113) | ABT-888 20 mg BID + TMZ QD (N=116) | ABT-888 40 mg BID + TMZ QD (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 9 | 19 | 13
LEUKOPENIA (Blood and lymphatic system disorders) | 5 | 8 | 8
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 | 4 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 24 | 26
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 19 | 49 | 56
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 11 | 15
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 4 | 6
CONSTIPATION (Gastrointestinal disorders) | 62 | 60 | 62
DIARRHOEA (Gastrointestinal disorders) | 24 | 27 | 26
DRY MOUTH (Gastrointestinal disorders) | 6 | 3 | 0
DYSPEPSIA (Gastrointestinal disorders) | 12 | 8 | 8
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 10 | 2
NAUSEA (Gastrointestinal disorders) | 75 | 83 | 82
VOMITING (Gastrointestinal disorders) | 53 | 42 | 30
CHEST PAIN (General disorders) | 4 | 5 | 6
CHILLS (General disorders) | 4 | 8 | 8
FATIGUE (General disorders) | 73 | 75 | 77
INFLUENZA LIKE ILLNESS (General disorders) | 4 | 6 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 9 | 4
PAIN (General disorders) | 8 | 10 | 12
PYREXIA (General disorders) | 6 | 7 | 4
SINUSITIS (Infections and infestations) | 5 | 7 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 8 | 10
HAEMOGLOBIN DECREASED (Investigations) | 6 | 3 | 3
PLATELET COUNT DECREASED (Investigations) | 4 | 12 | 10
WEIGHT DECREASED (Investigations) | 7 | 7 | 6
DECREASED APPETITE (Metabolism and nutrition disorders) | 37 | 26 | 36
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 | 4 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 17 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 21 | 14
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 | 7 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 11 | 11 | 9
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 | 4 | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 13 | 10
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 6
DIZZINESS (Nervous system disorders) | 17 | 19 | 15
DYSGEUSIA (Nervous system disorders) | 8 | 15 | 11
HEADACHE (Nervous system disorders) | 30 | 22 | 25
LETHARGY (Nervous system disorders) | 7 | 6 | 6
ANXIETY (Psychiatric disorders) | 7 | 6 | 5
INSOMNIA (Psychiatric disorders) | 12 | 12 | 14
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 28 | 18
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 | 17 | 17
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 10
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 5
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 | 2 | 8
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 7 | 3
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 | 3 | 2
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 7 | 7 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 7 | 6
RASH (Skin and subcutaneous tissue disorders) | 6 | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.